CLINICAL TRIAL: NCT03821636
Title: Impact of Long Alimentary Limb or Long Biliary Limb Roux-en-Y Gastric Bypass on Type 2 Diabetes Remission in Severely Obese Patients. A Prospective, Multicentric, Randomized, Controlled Trial.
Brief Title: Impact of Long Alimentary Limb or Long Biliary Limb Roux-en-Y Gastric Bypass on Type 2 Diabetes Remission in Severely Obese Patients.
Acronym: PRECI-Surg
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017_02; 2017-A01761-52 (Other: ID-RCB number, ANSM); PHRCI-16-090 (Other: PHRC number, DGOS)
Record Dates: First submitted 2018-11-26; First posted 2019-01-30 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus Type 2 in Obese
Keywords: Obesity; Diabetes Mellitus Type 2; Bariatric Surgery; Roux-en-Y; gastric bypass
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Roux-en-Y (Sham Comparator)
  Interventions: Procedure: Standard Roux-en-Y gastric bypass
- Long alimentary limb Roux-en-Y (Active Comparator)
  Interventions: Procedure: Long alimentary limb Roux-en-Y gastric bypass

INTERVENTIONS:
Procedure: Standard Roux-en-Y gastric bypass — Standard Roux-en-Y gastric bypass is performed with a 30 ml gastric pouch, a stapled gastrojejunal anastomosis with an alimentary limb of 25 % of total length of the intestine (150 cm), connected to the biliary limb of 10 % of total length of the intestine (60 cm) below the duodeno-jejunal junction with a side-to-side jejuno-jejunal anastomosis and a common limb of 65 % of total length of the intestine (400 cm).
  Arms: Standard Roux-en-Y
Procedure: Long alimentary limb Roux-en-Y gastric bypass — Long alimentary limb Roux-en-Y gastric bypass is performed with a 30 ml gastric pouch, a stapled gastrojejunal anastomosis with an alimentary limb of 45 % of total length of the intestine (280 cm), connected to the biliary limb of 10 % of total length of the intestine (60 cm) below the duodeno-jejunal junction with a side-to-side jejuno-jejunal anastomosis and a common limb of 45 % of total length of the intestine (280 cm
  Arms: Long alimentary limb Roux-en-Y

SUMMARY:
In patients with type 2 diabetes, Roux-en-Y gastric bypass (RYGB), which excludes a portion of the stomach and the proximal intestine from the alimentary circuit, improves glucose metabolism more rapidly and more extensively than is expected from weight loss. The mechanisms of this unique effect of gastrointestinal exclusion appear to be complex and have not yet been clarified. A recent study unveil that intestinal uptake of ingested glucose is diminished by RYGB and restricted to the common limb, where food meets bile and other digestive fluids, resulting in an overall decrease of post prandial blood glucose excursion. the hypothesize that reducing the length of the common limb, which is rarely measured and highly variable in clinical practice, may significantly affect the metabolic outcome of gastrointestinal surgical procedures. The aim of the present study is to compare the impact of two variants of Roux-en-Y gastric bypass with a short common limb, the long alimentary limb or the long biliary limb Roux-en-Y gastric bypass, on type 2 diabetes remission in severely obese patients.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 35 kg/m2
* All patient with type 2 diabetes
* Patients who were candidates for obesity surgery in accordance with French recommendation

Exclusion Criteria:

* Severe cognitive or mental disorders
* patient who have already undergone obesity surgery
* Severe and non-stabilised eating disorders
* The likely inability of the patient to participate in lifelong medical follow-up
* Alcohol or psychoactive substances dependence
* The absence of identified prior medical management of obesity
* Diseases that are life-threatening in the short and medium term;
* Contraindications to general anaesthesia.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 396 (Estimated)
Dates: Start 2019-06-16 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Rate of type 2 diabetes remission | at 12 months after surgery
  HbA1c < 6.5% AND fasting blood glucose < 7.0 mmol/L in absence of antidiabetic drug

SECONDARY OUTCOMES:
Absolute weight loss (aWL in kg) | at 1, 3, 6 and 12 months after surgery
Excess Weight Loss percentage (EWL%) | at 1, 3, 6 and 12 months after surgery
Excess BMI Loss percentage (EBL%) | at 1, 3, 6 and 12 months after surgery
Medical and surgical complication rates | During the month following surgery (for early complications) and from one month to 12 months postoperatively (for late complications)]
  Medical and surgical complication rates (anastomotic leaks, biliary reflux, bowel obstruction, anastomotic ulcers, anastomotic stenosis, internal hernia, chronic gastritis, esophagitis, iron deficiency anemia)
Type and severity of early and late complications for each procedure | During the month following surgery (for early complications) and from one month to 12 months postoperatively (for late complications)]
  Type and severity of early and late complications for each procedure, according to the Dindo-Clavien classification
Patient's quality of life score according to the Impact of Weight on Quality of Life (IWQOL) questionnaire | Before surgery and at 12 after surgery
  The IWQOL questionnaire to be specifically assess the effects of obesity on health-related quality of life. The five identified scales are Physical Function, Self-Esteem, Sexual Life, Public Distress, and Work.
  The final 20-item IWQOL includes two primary domains: Physical (7 items) and Psychosocial (13 items)
Patient's quality of life score according to the Gastrointestinal Quality of Life Index (GIQLI) questionnaire adapted to bariatric surgery. | Before surgery and at 12 after surgery
  GIQLI (gastrointestinal quality of life index) questionnaire. 36 questions, each containing 4 answers equating to a score ranging from 0 (least desirable answer) to 4 (most desirable answer). Total score range 0-144.
Change in glucose homeostasis | Before surgery and at 3, 6 and 12 months after surgery
  glucose (mg/dl)
Change in HbA1c | Before surgery and at 3, 6 and 12 months after surgery
  Changes in HbA1c(%) were assessed before and after surgery
Change in fasting glycemia | Before surgery and at 3, 6 and 12 months after surgery
  Changes in fasting blood glucose levels (mmol/L)
changes in fasting insulinemia | Before surgery and at 3, 6 and 12 months after surgery
  Changes in fasting insulinemia in microunits/mL
change in fasting c-peptide | Before surgery and at 3, 6 and 12 months after surgery
  Changes in C-peptide(ng/ml) were assessed before and after the intervention.
Number of antidiabetic treatments | Before surgery and at 3, 6 and 12 months after surgery
  Metabolic profile of glucose homeostasis assessment according to antidiabetic treatments, HbA1c level, fasting glycemia, fasting insulinemia fasting c-peptide
Changes in blood lipids profile | Before surgery and at 1, 3, 6 and 12 months after surgery
  Changes in blood lipids profile (LDL, HDL and triglyceride concentrations) according to anitilipidemic treatments
change in vitamins status assessment | Before surgery and at 1, 3, 6 and 12 months after surgery
  vitamines profil (vitamin B1, B9, B12, and D concentration) before and 12 and 24 months after surgery
change in prealbumin levels | Before surgery and at 1, 3, 6 and 12 months after surgery
  Lower levels of prealbumin are associated with malnutrition.

CONTACTS AND LOCATIONS:
Overall Officials: Grégory BAUD, MD, Principal Investigator — University Hospital, Lille
Locations (4):
- France (4):
  - Chu Amiens Picardie, Amiens
  - Ch Boulogne-Sur-Me, Boulogne-sur-Mer
  - Hop Claude Huriez Chu Lille, Lille
  - Ch de Valenciennes, Valenciennes